CLINICAL TRIAL: NCT04081116
Title: The Optimal Settings of MI-E in Children With NMD and Weak Cough
Brief Title: Mechanical Insufflation -Exsufflation in Children With NMD and Weak Cough
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Brit Hov, Physiotherapist, Oslo University Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18/12375
Record Dates: First submitted 2019-02-04; First posted 2019-09-09 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Neuromuscular Diseases in Children

STUDY DESIGN:
Intervention Model Description: Three different settings are tested on the same patients but in randomized order.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, care provider, investigator and outcomes assessor are blinded from the order of the settings tested. Only a technician change settings and know the order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MI-E testing symmetric settings (Experimental): Symmetric settings is one of 3 different settings that will be tested on the same day but in randomized order.
  Interventions: Other: Symmetric settings (high pressures/fast rate); Other: Asymmetric settings (Pi<Pe/Ti>Te); Other: Preinclusion settings
- MI-E testing assymetric settings (Experimental): Asymmetric settings is one of 3 different settings that will be tested on the same day but in randomized order.
  Interventions: Other: Symmetric settings (high pressures/fast rate); Other: Asymmetric settings (Pi<Pe/Ti>Te); Other: Preinclusion settings
- Settings in use (Sham Comparator): Settings in use is one of 3 different settings that will be tested on the same day but in randomized order
  Interventions: Other: Symmetric settings (high pressures/fast rate); Other: Asymmetric settings (Pi<Pe/Ti>Te); Other: Preinclusion settings

INTERVENTIONS:
Other: Symmetric settings (high pressures/fast rate) — Describes settings on the MI-E device
Other: Asymmetric settings (Pi<Pe/Ti>Te) — Lower insufflation pressures at longer times
Other: Preinclusion settings — Settings in use at start of study

SUMMARY:
Neuromuscular diseases (NMD) in children are severe, possibly life-threatening orphan conditions. The children are vulnerable and often subject to rapid deterioration of pulmonary function due to impaired ability to clear airway secretions. The use of mechanical cough augmentation with insufflation-exsufflation (MIE) is a strategy to treat and prevent. Possible major benefits are described, but optimal settings for best efficacy and comfort in children are not established. The project aim to improve the quality of the treatment with MIE in children with NMD and weak cough. On the basis of a bench study a clinical trial aims to examine the most effective MIE settings when used in stable state and when respiratory tract infections are present.

DETAILED DESCRIPTION:
On the basis of a prevalence study and a bench study different settings will be studied in children with NMD and weak cough to examine if settings derived from the lung model, are optimal to increase the peak cough flow (PCF) and comfort measured by visual analogue scale (VAS) in children with NMD and weak cough.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed neuromuscular disease < 18 years
* Established use (> 3mnd) of MI-E.
* Reduced PCF

  * PCF < 270 l/min (when > 12 years)
  * < 5th percentiles for PCF 16 (when 4 - 12 years)
* Clinical indication (difficulty to clear secretions, audible weak cough, history of pneumonia or frequent or prolonged respiratory tract infections).

Exclusion Criteria:

* age < 6 mnd
* obstructive lung disease (hyperinflation or emphysema on x-ray.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 77 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
PCF in the MI-E circuit | 30 minutes.
  Recording of maximal value produced by the MI-E device during Cough
Patient reported comfort | Total time use 30 min
  Comfort rated on a Visual Analog Scale (VAS) (0-100) where 100 is very uncomfortable and 0 is very comfortable.

SECONDARY OUTCOMES:
Carbon dioxide | maximal time use is 30 min
  Transcutaneous trend measurement of CO2 during data collection
Oxygen | maximal time use is 30 min
  Transcutaneous trend measurement of peripheral O2 during data collection
Hart rate | Total max 30 minutes (During three MI-E trials)
  Transcutaneous trend measurement of hart rate during data collection
Patient reported efficacy | The VAS is recorded after each of the three trials. Total time use 30 min
  Efficacy rated on a Visual Analog Scale (0-100) where 100 is not efficient at all and 0 is very efficient.

CONTACTS AND LOCATIONS:
Locations (4):
- Norway (4):
  - Helse bergen HF, Bergen
  - Oslo university hospital, Oslo
  - Stavanger university hospital, Stavanger
  - St. Olav Trondheim university hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morrow B, Argent A, Zampoli M, Human A, Corten L, Toussaint M. Cough augmentation techniques for people with chronic neuromuscular disorders. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013170. doi: 10.1002/14651858.CD013170.pub2. PMID 33887060